CLINICAL TRIAL: NCT00486668
Title: A Randomized Phase III Trial of Neoadjuvant Therapy for Patients With Palpable and Operable HER2-Positive Breast Cancer Comparing the Combination of Trastuzumab Plus Lapatinib to Trastuzumab and to Lapatinib Administered With Weekly Paclitaxel Following AC Accompanied by Correlative Science Studies to Identify Predictors of Pathologic Complete Response
Brief Title: A Study of AC Followed by a Combination of Paclitaxel Plus Trastuzumab or Lapatinib or Both Given Before Surgery to Patients With Operable HER2 Positive Invasive Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-41
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Invasive Breast Cancer
Keywords: HER2 positive breast cancer; invasive breast cancer; lapatinib; neoadjuvant; NSABP; paclitaxel; trastuzumab; doxorubicin; cyclophosphamide
MeSH Terms: interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; Trastuzumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: AC then paclitaxel + trastuzumab (Active Comparator): AC followed by paclitaxel plus trastuzumab
  Interventions: Drug: doxorubicin; Drug: cyclophosphamide; Drug: paclitaxel; Drug: trastuzumab
- Group 2: AC then paclitaxel + lapatinib (Experimental): AC followed by paclitaxel plus lapatinib
  Interventions: Drug: doxorubicin; Drug: cyclophosphamide; Drug: paclitaxel; Drug: lapatinib
- Group 3: AC then paclitaxel + trastuzumab + lapatinib (Experimental): AC followed by paclitaxel plus trastuzumab plus lapatinib
  Interventions: Drug: doxorubicin; Drug: cyclophosphamide; Drug: paclitaxel; Drug: trastuzumab; Drug: lapatinib

INTERVENTIONS:
Drug: doxorubicin — 60 mg/m2 IV every 21 days for cycles 1-4
Drug: cyclophosphamide — 600 mg/m2 IV every 21 days for cycles 1-4
Drug: paclitaxel — 80 mg/m2 IV on days 1, 8, and 15 every 28 days for cycles 5-8
Drug: trastuzumab — First dose: 4 mg/kg IV, subsequent doses: 2 mg/kg IV weekly beginning on day 1 of the first paclitaxel cycle until 1-7 days before surgery
  Arms: Group 1: AC then paclitaxel + trastuzumab; Group 3: AC then paclitaxel + trastuzumab + lapatinib
Drug: lapatinib — Group 2: 1250 mg PO daily beginning on day 1 of the first paclitaxel cycle until 1 day before surgery. Group 3: 750 mg PO daily beginning on day 1 of the first paclitaxel cycle until 1 day before surgery.
  Arms: Group 2: AC then paclitaxel + lapatinib; Group 3: AC then paclitaxel + trastuzumab + lapatinib

SUMMARY:
The primary purpose of this study is to determine whether breast cancer tumors respond (as measured by pathologic complete response: the absence of microscopic evidence of invasive tumor cells in the breast) to combined chemotherapy of AC(doxorubicin and cyclophosphamide) followed by paclitaxel plus trastuzumab or lapatinib or both given before surgery to patients with HER2-positive breast cancer. Trastuzumab will also be given to all patients after surgery. The study will also evaluate the toxic effects of the chemotherapy combination, including effects on the heart, and will determine survival and progression-free survival 5 years after treatment. Also, the study will look at whether there are gene expression profiles in the tumor tissue that can predict pathologic complete response.

DETAILED DESCRIPTION:
Women with breast cancers that overexpress HER2 are at greater risk for disease progression and death than women whose tumors do not overexpress HER2. Trastuzumab, a recombinant humanized monoclonal antibody against the extracellular domain of the HER2 protein blocks downstream signaling of HER2 and substantially improves the efficacy of chemotherapy in women with metastatic and early-stage HER2-positive breast cancers. Because resistance to trastuzumab eventually results in progressive disease in the metastatic setting and contributes to recurrence following adjuvant trastuzumab-based therapy, it is important to develop agents other than trastuzumab that target HER2 signaling through different mechanisms of action. Lapatinib is an oral, small molecule, dual tyrosine kinase inhibitor of HER2 and EGFR. Lapatinib has shown a lack of cross-resistance with trastuzumab in preclinical studies and activity in women with HER2-positive, metastatic breast cancer that has progressed during trastuzumab treatment. Trastuzumab blocks the downstream signaling of HER2 by binding to the extracellular domain of the receptor. Lapatinib binds to the intracellular domains of HER2 and EGFR and prevents activation of downstream signaling pathways. Because of this different mechanism of action, lapatinib may be effective in trastuzumab-resistant disease. The study will also provide important safety information on trastuzumab and lapatinib combinations immediately following anthracycline exposure, and also provide an initial direct comparison of cardiac effects of trastuzumab and lapatinib when incorporated into a standard sequential AC followed by weekly paclitaxel (neo)adjuvant regimen.

Availability of a second agent that can interrupt HER2-signaling pathways through completely different mechanisms than those of trastuzumab offers the potential for further improvement in the management of patients with HER2-overexpressing breast cancer in both the adjuvant and metastatic setting. Co-administration of both trastuzumab and lapatinib with chemotherapy may be important in improving outcomes in subsets of HER2-positive breast cancers. However, use of two inhibitors of the HER2 pathway will increase costs and may increase toxicity, so it will be important to identify the subsets of patients who would benefit from the dual therapy. Inhibition of HER2 with a single agent clearly is sufficient for many patients as evidenced by the results of the trastuzumab trials. Therefore, co-administration to unselected populations of women with HER2-positive breast cancers would not represent an optimal approach. Given the activity of lapatinib, it is likely that it will also be sufficiently active in inhibiting HER2-pathway activation in some patients to allow for its use as the sole inhibitor of the HER2 pathway. Different populations may also derive greater benefit from one of the HER2-blocking agents relative to the other. Identification of potential predictive factors for pathologic complete response to the combination or to either agent administered alone in neoadjuvant trials would provide important information for adjuvant trials designed to definitively address these important issues.

This study will compare 3 combined chemotherapy regimens: AC followed by paclitaxel plus trastuzumab and lapatinib, AC followed by paclitaxel plus lapatinib, and AC followed by paclitaxel plus trastuzumab given before surgery to patients with HER2-positive breast cancer.

ELIGIBILITY:
Inclusion criteria:

* Female
* 18 years or older
* ECOG performance status of 0 or 1
* Primary breast tumor palpable and measures greater than or equal to 2.0 cm by physical exam
* Diagnosis of invasive adenocarcinoma made by core needle biopsy
* Breast cancer determined to be HER2-positive
* LVEF assessment by MUGA scan or ECG within 3 months prior to randomization
* Blood counts must meet the following criteria:

  * ANC greater than or equal to 1200/mm3
  * Platelet count greater than or equal to 100,000/mm3
  * Hemoglobin greater than or equal to 10 g/dL
* Serum creatinine less than or equal to ULN for the lab
* Adequate hepatic function by these criteria:

  * Total bilirubin less than or equal to the ULN for the lab unless the patient has a bilirubin elevation greater than ULN to 1.5 x ULN resulting from Gilbert's disease or similar syndrome due to slow conjugation of bilirubin; and
  * Alkaline phosphatase less than or equal to 2.5 x ULN; and
  * AST less than or equal to 1.5 x ULN for the lab.
* If skeletal pain present or alkaline phosphatase greater than ULN (but less than or equal to 2.5 x ULN), bone scan or PET scan must not demonstrate metastatic disease
* If AST or alkaline phosphatase greater than ULN , liver imaging (CT, MRI or PET scan) must not demonstrate definitive metastatic disease and the requirements in criterion for hepatic function must be met
* Able to swallow oral medications

Exclusion criteria:

* FNA alone to diagnose the primary tumor
* Excisional biopsy or lumpectomy was performed prior to randomization
* Surgical axillary staging procedure prior to randomization. Exceptions: 1) FNA or core biopsy of an axillary node for any patient, and 2) although not recommended, a pre-neoadjuvant therapy SN biopsy for patients with clinically negative axillary nodes.
* Tumors clinically staged as T4
* Ipsilateral cN2b or cN3 disease (Patients with cN1 or cN2a disease are eligible)
* Definitive clinical or radiologic evidence of metastatic disease
* Synchronous bilateral invasive breast cancer
* Requirement for chronic use of any of the medications or substances specified in the protocol
* Treatment including RT, chemotherapy, and/or targeted therapy for the currently diagnosed breast cancer prior to randomization
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormone replacement therapy, etc. (These patients are eligible if therapy is discontinued prior to randomization)
* Continued therapy with any hormonal agent such as raloxifene, tamoxifen, or other SERM. (Patients are eligible only if these medications are discontinued prior to randomization)
* Prior history of breast cancer, including DCIS (Patients with a history of LCIS are eligible)
* Prior therapy with anthracyclines, taxanes, trastuzumab, or lapatinib for any malignancy
* Other malignancies unless the patient is considered to be disease-free for 5 or more years prior to randomization and is deemed by her physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Cardiac disease that would preclude the use of the drugs included in the B-41 treatment regimens. This includes but is not confined to:

  * Active cardiac disease:

    * angina pectoris requiring the use of anti-anginal medication;
    * ventricular arrhythmias except for benign premature ventricular contractions controlled by medication;
    * conduction abnormality requiring a pacemaker;
    * supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; and
    * clinically significant valvular disease.
  * History of cardiac disease:

    * myocardial infarction;
    * congestive heart failure; or
    * cardiomyopathy.
* Uncontrolled hypertension, defined as blood pressure greater than 150/90 mm/Hg on antihypertensive therapy
* History of or current symptomatic interstitial pneumonitis or pulmonary fibrosis or definitive evidence of interstitial pneumonitis or pulmonary fibrosis described on CT or chest x-ray in asymptomatic patients
* Sensory/motor neuropathy greater than or equal to grade 2, as defined by the NCI's CTCAE v3.0
* Malabsorption syndrome, ulcerative colitis, resection of the stomach or small bowel, or other disease significantly affecting gastrointestinal function
* Other non-malignant systemic disease that would preclude treatment with any of the treatment regimens or would prevent required follow-up
* Conditions that would prohibit administration of corticosteroids
* Administration of any investigational agents within 30 days before randomization
* Pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2007-07; Primary Completion 2012-06 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Determination of pathologic complete response (pCR), defined by the absence of microscopic evidence of invasive tumor cells in the post chemotherapy surgical breast specimen. | surgery following chemotherapy

SECONDARY OUTCOMES:
The determination of pCR in the surgical breast and lymph node specimens following chemotherapy. | surgery following chemotherapy
Clinical tumor measurement as assessed by physical exam of the breast and lymph nodes | baseline (prior to starting protocol therapy), at the completion of AC (before starting paclitaxel and trastuzumab and/or lapatinib), and at the conclusion of the sequential regimens (prior to surgery).
Determination of cardiac toxicity as measured by the incidence of cardiac events defined as definite or probable cardiac death | two year cumulative incidence
Determination of non-cardiac toxicities as measured by frequencies of adverse events categorized using CTCAE v3.0. | through 5 years after entry
Overall survival as measured by time from randomization until death from any cause. | through 5 years after entry
Recurrence-free interval as measured by occurrence of inoperable progressive disease, or from time of surgery to occurrence of local, regional, or distant recurrence in patients with operable disease. | through 5 years after entry
In tumor tissue, a comparison of array comparative genomic hybridization (CGH) data with gene expression profile data to examine coordinated overexpression of amplified genes, especially in HER2 and cMYC loci. | Tissue sample collected at surgery following chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (110):
- United States (103):
  - MBCCOP, Gulf Coast, Mobile, Alabama
  - Scripps Cancer Center-San Diego, La Jolla, California
  - University of California, Irvine Medical Center, Long Beach, California
  - Pacific Shores Medical Group, Long Beach, California
  - St. Joseph Hospital, Orange, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Stanford University Medical Center, Palo Alto, California
  - Sutter Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego, San Diego, California
  - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Memorial Hospital, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - CCOP-Colorado Cancer Research Prog. Inc.(Administrative Only), Denver, Colorado
  - Kaiser Permanente Rock Creek, Lafayette, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Eastern Connecticut Hematology & Oncology Associates, Norwich, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - MD Anderson Cancer Center, Orlando, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - MBCCOP, Medical College of Georgia Research Institute, Augusta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Kaiser Permanente Hawaii - Moanalua Med Center, Honolulu, Hawaii
  - Kootenai Cancer Center, Coeur d'Alene, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Cancer Institute at Alexian Brothers Hospital Network, Elk Grove, Illinois
  - Edward Hospital, Naperville, Illinois
  - Edward Cancer Center Plainfield, Plainfield, Illinois
  - CCOP, Central Illinois, Springfield, Illinois
  - CCOP, Carle Cancer Center, Urbana, Illinois
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - CCOP, Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - CCOP, Des Moines, IA, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa
  - CCOP, Sioux Community Cancer consortium, Sioux City, Iowa
  - CCOP, Wichita KS, Wichita, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - NortonHealtcare Inc., Louisville, Kentucky
  - CCOP, Ochsner Clinic Foundation, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - CCOP, Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP, Grand Rapids Clnical Oncology Program, Grand Rapids, Michigan
  - CCOP, Kalamazoo, MI, Kalamazoo, Michigan
  - Michigan State University - Breslin Cancer Center, Lansing, Michigan
  - CCOP, William Beaumont Hospital, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - CCOP, Metro-Minnesota, Minneapolis, Minnesota
  - University of Missouri-Ellis Fischel, Columbia, Missouri
  - CCOP, Kansas City (Administrative Only), Kansas City, Missouri
  - CCOP, Ozark Health Ventures LLC, Springfield, Missouri
  - Saint Louis UniversityHealth Sciences Center, St Louis, Missouri
  - CCOP, Heartland Cancer Research, St Louis, Missouri
  - CCOP, Montana Cancer Consortium, Billings, Montana
  - CCOP, Missouri Valley Consortium, Omaha, Nebraska
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York Oncology Hematology PC-Albany, Albany, New York
  - Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - CCOP, Hematology-Oncology Associates of CNY, Syracuse, New York
  - Alamance Regional Medical Center, Burlington, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - CCOP, Southeast Cancer Control Consortium, Charlotte, North Carolina
  - Alamance Regional Medical Center - Off site Clinic, Mebane, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Aultman Hospital, Canton, Ohio
  - Case Western Reserve/University Hospitals-Ireland Cancer Cntr., Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - CCOP, Columbus, OH, Columbus, Ohio
  - CCOP, Dayton, OH, Dayton, Ohio
  - CCOP, Oklahoma, Tulsa, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Clinic, Danville, Pennsylvania
  - Hershey Medical Center, Hershey, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Allegheny General Hospital/Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - NSABP Foundation, Inc., Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Reading Hospital & Medical Center, West Reading, Pennsylvania
  - CCOP, Main Line Health, Wynnewood, Pennsylvania
  - CCOP, Upstate Carolina, Spartanburg, South Carolina
  - Sanford Cancer Center, Souix Falls, South Dakota
  - Thompson Cancer Survival Center-Dowell Springs, Knoxville, Tennessee
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP, Virginia Commonwealth University, Richmond, Virginia
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP, Virginia Mason, Seattle, Washington
  - CCOP, Northwest, Tacoma, Washington
  - West Virginia University Hospitals Inc., Morgantown, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - CCOP, Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - Odette Cancer Centre, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - University of Montreal Hospital Group, Montreal, Quebec
  - Centre Hospitalier Affilie Universitaire De Quebec, Hospital du St-Sacrement, Québec, Quebec
- MBCCOP, San Juan, Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Robidoux A, Tang G, Rastogi P, Geyer CE Jr, Azar CA, Atkins JN, Fehrenbacher L, Bear HD, Baez-Diaz L, Sarwar S, Margolese RG, Farrar WB, Brufsky AM, Shibata HR, Bandos H, Paik S, Costantino JP, Swain SM, Mamounas EP, Wolmark N. Lapatinib as a component of neoadjuvant therapy for HER2-positive operable breast cancer (NSABP protocol B-41): an open-label, randomised phase 3 trial. Lancet Oncol. 2013 Nov;14(12):1183-92. doi: 10.1016/S1470-2045(13)70411-X. Epub 2013 Oct 4. PMID 24095300
- [Derived] Rastogi P, Tang G, Hassan S, Geyer CE Jr, Azar CA, Magrinat GC, Suga JM, Bear HD, Baez-Diaz L, Sarwar S, Boileau JF, Brufsky AM, Shibata HR, Bandos H, Paik S, Yothers G, Swain SM, Mamounas EP, Wolmark N. Long-term outcomes of dual vs single HER2-directed neoadjuvant therapy in NSABP B-41. Breast Cancer Res Treat. 2023 Jun;199(2):243-252. doi: 10.1007/s10549-023-06881-8. Epub 2023 Mar 22. PMID 36944848